CLINICAL TRIAL: NCT02752984
Title: Prospective Study on the Incidence of Early Deep Vein Thrombosis After Peripherally Inserted Central Catheter Insertion
Brief Title: Study on the Incidence of Early Deep Vein Thrombosis After Peripherally Inserted Central Catheter Insertion
Acronym: DVT-PICC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Michele Pagani, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: TROMBOSI VENOSA PROFONDA
Record Dates: First submitted 2016-04-11; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Venous Thrombosis
Keywords: Peripherally inserted central venous catheter
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PICC insertion: Peripherally Inserted Central Catheter insertion

SUMMARY:
Deep Vein Thrombosis (DVT) is one of the most important complications after Peripherally Inserted Central Catheter (PICC) insertion. This study goals are to understand when and why DVT develops.

DETAILED DESCRIPTION:
Deep Vein Thrombosis (DVT) is one of the most important complications after Peripherally Inserted Central Catheter (PICC) insertion. This study goals are to understand when and why DVT develops. Patients will be studied with ultrasound for 4 weeks after PICC insertion, one visit a week. The final outcome of PICCs will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Peripherally Inserted Central Catheter insertion

Exclusion Criteria:

* Pre-existing Deep Vein Thrombosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with Peripherally Inserted Central Catheter insertion
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Early Deep Vein Thrombosis incidence assessed with weekly ultrasound examination | 4 weeks

SECONDARY OUTCOMES:
Factors which may be correlated to Deep Vein Thrombosis development: obesity (Body Mass Index) | 4 weeks
  Body Mass Index (kg/m^2)
Factors which may be correlated to Deep Vein Thrombosis development: cancer | 4 weeks
  Cancer yes/no
Factors which may be correlated to Deep Vein Thrombosis development: previous Deep Vein Thrombosis | 4 weeks
  Previous Deep Vein Thrombosis yes/no
Factors which may be correlated to Deep Vein Thrombosis development: Heparin-induced thrombocytopenia | 4 weeks
  Heparin-induced thrombocytopenia yes/no
Overall Deep Vein Thrombosis incidence | 6 months
  Number of patients with Deep Vein Thrombosis/total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Michele Pagani, MD, Principal Investigator — IRCCS Policlinico San Matteo Pavia
Locations (1):
- IRCCS Policlinico San Matteo Pavia, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chopra V, Ratz D, Kuhn L, Lopus T, Lee A, Krein S. Peripherally inserted central catheter-related deep vein thrombosis: contemporary patterns and predictors. J Thromb Haemost. 2014 Jun;12(6):847-54. doi: 10.1111/jth.12549. PMID 24612469
- [Background] Zochios V, Umar I, Simpson N, Jones N. Peripherally inserted central catheter (PICC)-related thrombosis in critically ill patients. J Vasc Access. 2014 Sep-Oct;15(5):329-37. doi: 10.5301/jva.5000239. Epub 2014 Apr 25. PMID 24811591